CLINICAL TRIAL: NCT00001070
Title: A Dose Escalation Study to Evaluate Tolerance and Antiviral Effect of Oral Vitamin C in Two Groups of HIV-Infected Adults
Brief Title: The Safety and Effectiveness of Different Doses of Vitamin C in HIV-Infected Patients
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Purpose: Treatment
Other Study IDs: DATRI 017
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2023-04-14 (Actual); Status verified 2023-04

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections | interventions — Ascorbic Acid

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Oral Vitamin C

SUMMARY:
This is a study to evaluate the tolerance and antiviral effect of oral vitamin C in HIV-infected.

ELIGIBILITY:
Not applicable - Study withdrawn since 04/23/1996

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)